CLINICAL TRIAL: NCT07332182
Title: Multicenter Prospective Randomized Study of MaioRegenTM Prime vs. Debridement (Surgical Standard of Care (SSOC)) for the Treatment of Osteochondral Lesion of the Knee Joint - OSTEOCONFIRM Study
Brief Title: MaioRegen Prime Study for the Treatment of Deep Osteochondral Lesion of the Knee
Acronym: OSTEOCONFIRM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fin-Ceramica Faenza Spa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORT-24
Record Dates: First submitted 2026-01-07; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Osteochondral Lesions of the Knee Joint; Osteochondritis Dissecans (OCD); Early Osteoarthritis
Keywords: osteochondral lesion; MaioRegen Prime; OCD; knee; scaffold; biomimetic
MeSH Terms: conditions — Osteochondritis Dissecans; Osteoarthritis

STUDY DESIGN:
Masking Description: CEC (clinical event committee) board members will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MaioRegen Prime (Experimental): Medical Device: MaioRegen Prime implant
  Interventions: Device: osteochondral scaffold implant
- Surgical Standard of Care (SSOC) (Active Comparator): Debridement
  Interventions: Procedure: SSOC

INTERVENTIONS:
Device: osteochondral scaffold implant — three layered biomimetic osteochondral scaffold implant for osteochondral lesions of the knee
  Arms: MaioRegen Prime
Procedure: SSOC — Debridement
  Arms: Surgical Standard of Care (SSOC)

SUMMARY:
The present study aims to compare the efficacy and the safety of MaioRegen Prime to Debridement (SSOC) in patients with deep osteochondral lesions of the knee joint. The foreseen population involves patients with osteochondral lesions with different etiology, dimension, shape, and location.

The evaluation will be performed through clinical, subjective and objective assessments.

DETAILED DESCRIPTION:
This is multicenter, prospective, randomized clinical trial, subjects will be randomized (2:1) to MaioRegen Prime or debridement.

All randomized patients will be followed with post-operative visits at 15 days, 6 weeks, 3, 6, 12, 18 and 24 months after surgery and annually post-24 months visit (until last patient reaches 24 months).

During screening period and at follow-up visits commonly used specific scores will be evaluated: IKDC Subjective Knee Evaluation Form, IKDC Knee Examination Form, KOOS, Tegner Score, VAS pain, PROMIS-29, ICRS Cartilage Repair Assessment and MRI related scores.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent prior to any study-related procedures;
2. Male or female patients aged between 18 and 60 years (inclusive);
3. Body Mass Index (BMI) ≤ 35;
4. Up to 3 treatable osteochondral lesions localized in femoral condyles and/or trochlea (the patient might have other lesion in other parts of the joint, but they should not be more severe than ICRS Grade II lesions as determined by baseline MRI);
5. Knee osteochondral lesion(s) (Grade IVa and IVb according to ICRS Classification) or not re-fixable knee Osteochondritis Dissecans lesions as determined by baseline MRI;
6. Lesions with an overall treatable area 1-7 cm2 (as determined by baseline MRI). In case of multiple lesions (maximum 3 lesions) in the same knee compartment a minimum distance of 3 mm is required);
7. IKDC Subjective score at baseline (pre-op evaluation) is less than 70;
8. Non-responsive to physical therapy for at least 6 weeks;
9. Patients physically and mentally willing and able to comply with the post-operative rehabilitation protocol and scheduled clinical and radiographic visits.

Exclusion Criteria:

1. IKDC subjective score at Baseline is more than or equal to 70;
2. KOOS Pain Subscale score at baseline is less than 20 or more than 65 (scale: maximum pain = 0, pain free = 100);
3. Osteochondral tibial plateau and/or patella defects;
4. Patients affected by advanced osteoarthritis in the index knee (Kellgren and Lawrence classification 3 or 4);
5. Bony defect depth deeper than 5 mm, according to baseline MRI, measured from the original subchondral bone plate level;
6. Uncontained defects: lack of vital bone wall at least 2 mm thick, completely surrounding the lesion - based on MRI;
7. Patients with untreated patellofemoral malalignment or who have undergone realignment procedures within 6 months;
8. Patients with bone fracture or uncorrected malalignment more than 5 degrees varus or valgus according to standing X-ray.
9. Patients previously treated for total or partial meniscectomy in the specific index knee compartments (more than 50% of the meniscus in the index compartments is missing);
10. Patient requiring total or partial meniscectomy to be performed concomitantly, involving more than 50% of one or both menisci in the index knee compartment (lack of functional remaining meniscus, at least 5mm rim at the end of the procedure); and patient requiring ligamentoplasty and high tibial osteotomy (HTO) to be performed concomitantly;
11. Untreated knee ligament instability or treated within 6 months;
12. Kissing (counterposed) osteochondral lesions;
13. Significant instability of the index knee according to IKDC Knee Examination Form 2000: Grade C (abnormal) or D (severely abnormal).
14. Patients affected by any concomitant painful or disabling disease of the spine, hips, or lower limbs, including the contralateral knee, that would interfere with the evaluation of the index knee;
15. Patients affected by bilateral knee lesions that need treatment;
16. Intra-articular steroid injections within 3 months;
17. Any previous cartilage repair procedure (such as: microfracture, Osteochondral autograft transplantation system (OATS), Autologous Matrix Induced Chondrogenesis, (AMIC), Autologous Chondrocyte Implantation (ACI) with or without use of a scaffold (matrix) in the index knee within one year or debridement within 6 months;
18. Patients affected by osteoporosis (established through x-ray tests, called DEXA scans, bone density, etc. Criteria for osteoporosis: T-score is < - 2.5 SD), chondrodysplasia, or osteogenesis imperfecta;
19. Patients affected by known allergy to equine collagen or calcium-phosphates;
20. Patients who underwent chemotherapy in the past 12 months;
21. Patients with a known history of any significant systemic disease (such as but not limited to: HIV, hepatitis, HTLV, syphilis, coagulopathies, insulin dependent diabetes mellitus etc.) or affected by a significant malignancy;
22. Participation in other clinical trials within 90 days prior to the study or concurrent with the study;
23. Patient who is pregnant (or intends to become pregnant within one-year post-op) or breastfeeding;
24. Known drugs or alcohol abuse;
25. Any evidence of active infection anywhere in the body. Urinary Tract Infection (UTI) patients can be included following antibiotic treatment, and provided that two consecutive cultures are negative (taken within at least 2 weeks of each other);
26. Any known history of intra-articular or osseous infection of the index knee;
27. Patients affected by a known history of inflammatory arthropathy or crystal-deposition arthropathy;
28. Prisoners;
29. The existence of any surgical or medical condition that, in the judgement of the Investigator, might compromise patient safety or the outcome of the study;
30. Any medical conditions or implants that would prevent the participant from undergoing an MRI, including but not limited to pacemakers, clips, cochlear implants, or metal shrapnel.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Superiority of MaioRegen Prime vs Debridement | baseline, 24 months
  The primary endpoint is the success rate defined as a composite binary endpoint, where a patient is a success if they meet all of the following criteria:
  * At least a 15 points IKDC increase at 24 months
  * Lack of SAE related to MaioRegen treatment or debridement during the 24-month follow-up
  * Lack of related re-intervention after MaioRegen treatment or debridement during the 24-month follow-up

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score at 24 months of MaioRegen Prime compared to debridement | baseline, 24 months
  Subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function.
  The IKDC Subjective Knee Evaluation Form is graded by adding the results of each item's scores, and then converting the result to a scale from 0 to 100.
  Higher scores indicate higher levels of function and lower levels of symptoms, (i.e., a better outcome).
Rate of responder in IKDC Subjective Knee Evaluation at 24 months of MaioRegen Prime compared to debridement as defined as improvement in IKDC Subjective Knee Evaluation of ≥15 points | baseline, 24 months
  The new IKDC Subjective Knee Evaluation Form, published in 2000, is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function. The IKDC Subjective Knee Evaluation Form is graded by adding the results of each item's scores, and then converting the result to a scale from 0 to 100. Higher scores indicate higher levels of function and lower levels of symptoms, (i.e., a better outcome).
Proportion of patients without SAEs related to MaioRegen treatment or debridement treatment during the 24-month follow-up period | baseline, 24 months
Proportion of patients without related re-intervention after MaioRegen treatment or debridement treatment at 24 month follow-up period | baseline, 24 months
Change from baseline in average overall KOOS score (Knee Injury and Osteoarthritis Outcome Score) | baseline, 12, 18, and 24 months
  KOOS score consists of 5 subscales and covers: pain (9 items), symptoms (7 items, two of which are related to stiffness), functions and activities of daily living (17 items), physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items). Each question uses a 0 (no problem/difficulty) to 4 (extreme problem/difficulty) response, which is then converted into the final 0-100 score for each subscale, indicating the percentage of the total possible score achieved, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., better outcome).
Change from pre-injury and from baseline in Tegner score | baseline, 12 months, 18 months, 24 months
  Tegner activity level scale allows to know the level of physical activity carried out by the patients. Tegner's activity scale classifies the activity according to work and sports activities on a scale from 0 to 10, where 0 is being on sick leave/disabled due to knee issues, and 10 is elite, international competitive sports.
Change from baseline in IKDC (International Knee Documentation Committee) Knee Examination Objective Form | baseline, 12 months, 18 months, 24 months
  The IKDC objective examination form uses a 0-100 scale, calculated by summing seven parameters related to knee function. The presence of effusions and degree of knee motion are assessed; the worst value of any of these parameters determines the final IKDC grade. There are four grades (A, B, C, D) that identify a knee rated as normal, near normal, abnormal, and severely abnormal, respectively.
Change from baseline in VAS (visual analogue scale) pain | baseline, 12 months, 18 months, 24 months
  The VAS scale is a 0-cm line tool to measure pain intensity, with "no pain" at 0 and "worst pain imaginable" at 10, where patients mark their pain level
PROMIS-29 (Patient-Reported Outcomes Measurement Information System): Patient's QOL (quality of life) improvement | baseline, 12 months, 18 months and 24 months
  The PROMIS-29 uses a T-score metric (mean 50, SD 10) to assess 7 domains (Physical Function, Fatigue, Depression, Anxiety, Pain Interference, Sleep Disturbance, and Social Participation) with 4 questions with an additional pain intensity numeric rating scale (NRS, 0-10 score). There is no total score, but each axis forms its own score.
MRI evaluation: MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue) 2.0 Knee Score | baseline, 12 months, 24 months
  MOCART 2.0 score allows the assessment of both cartilage tissue repair and the structures surrounding it. It is a 0-100 point MRI-based system for evaluating cartilage repair, updating the original MOCART by focusing on nine key variables like defect filling (in 25% increments), integration to native cartilage, surface, signal intensity, bony changes (overgrowth/defect), marrow edema, and subchondral cysts. 100 represents the best score and a score of 0 represents the worst score.

OTHER OUTCOMES:
Safety Outcome | 24 monhs
  Adverse Events rate per type, severity, seriousness, and relatedness to the treatment, including Serious Adverse Events and Serious Adverse Device Effect, Adverse Device Effect, Unanticipated Adverse Device Effect, Re-operations, Complaint and Treatment Failures up to 24 months will be evaluated and adjudicated by CEC members.

IPD SHARING:
Plan to Share IPD: No